CLINICAL TRIAL: NCT06031064
Title: External Validation of a Clinical Scoring System to Predict Microscopic Colitis in Patients With Chronic Watery Diarrhoea
Brief Title: External Validation of a Microscopic Colitis Clinical Scoring System in Patients With Chronic Watery Diarrhoea
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Mutua de Terrassa (Other)
Responsible Party: Sponsor
Other Study IDs: P/22-108
Record Dates: First submitted 2023-08-28; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-08

CONDITIONS: Microscopic Colitis
Keywords: Inflammatory bowel disease (IBD); clinical scoring; chronic watery diarrhea
MeSH Terms: conditions — Colitis, Microscopic; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Frozen colon tissue and faecal sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic watery diarrhoea and clinical suspicion of MC

SUMMARY:
Chronic watery diarrhoea is a very common problem in the population and most of these patients will be referred for colonoscopy. If no macroscopic findings are observed during colonoscopy to justify the diarrhoea, serial colonic biopsies will be taken to rule out Microscopic Colitis (MC). However, it has been estimated that only 10-15% of these patients will be diagnosed with MC after colonoscopy. Therefore, about 80% of the biopsies collected and analysed will not be useful to establish a diagnosis, considerably increasing costs.

To predict the risk of developing MC, a new promising clinical scoring system has been recently developed. This score will be useful in the diagnostic work-up of chronic watery diarrhoea to prioritize colonoscopy with stepwise colonic biopsies in patients with a positive highly specific score for MC. In cases with a negative score, colonoscopy plus biopsies should be performed only if other diagnostic tests are negative.

The aim of this current study is to externally validate the new scoring system to predict MC in patients with chronic watery diarrhoea.

DETAILED DESCRIPTION:
Two diagnostic scoring systems have been proposed to predict the risk of developing MC: 1) The Kane score (sensitivity (SN) 96%; specificity (SP) 46%) combines eight risk factors, including female sex, age over 50 years, weight loss, absence of abdominal pain, and use of proton pump inhibitors (PPIs) and non-steroidal anti-inflammatory drugs (NSAIDs), presence of nocturnal diarrhoea and diarrhoea duration of less than 6 months. 2) The Cotter score (SN 93%; SP 49%) includes age ≥55 years, duration of diarrhoea ≤6 months, ≥5 bowel movements per day, body mass index <30 kg/m2, current smoking, and current use of selective serotonin reuptake inhibitors/serotonin-norepinephrine reuptake inhibitors and NSAIDs. However, both scoring systems have been derived from retrospective studies and watery chronic diarrhoea, the hallmark clinical symptom of MC, was not well defined.

Besides MC risk factors, faecal markers could also be useful for MC screening. Most studies have found that 60-75% of the patients with active collagenous colitis, a subtype of MC, have elevated faecal calprotectin levels. Moreover, a recent study showed that faecal calprotectin concentrations >100 μg/g (AUC, 0.73) showed a 67% sensitivity and 75% specificity to predict MC.

To further assess the value of the Kane and Cotter scoring systems and to derive a new score including faecal calprotectin aiming to increase specificity, the investigators performed a prospective observational two-centres study. Chronic watery diarrhoea was defined as ≥2 watery stools (Bristol 6-7) per day, of frequent occurrence (≥3 times per week), of at least 1 month duration. A registry of demographic and clinical characteristics (VAS of 0-100 of abdominal pain and abdominal distension, presence of nocturnal diarrhoea, urgency and faecal incontinence, smoking, body mass index, weight loss, use of drugs) was performed. The study included 118 patients with chronic watery diarrhoea, from which 41 were diagnosed with MC (21 lymphocytic colitis, 16 collagenous colitis and 4 paucicellular colitis) and obtained lower SN and SP values than those published of the Cotter (SN 78%; SP 57%) and Kane (SN 78%; SP 38%) scores. The AUC of both scores was 0.71 and 0.66, respectively. The multivariate analysis identified 5 variables associated with MC: >5 stools/day (OR 12.5), duration of diarrhoea ≤8 months (OR 5), regular use of low-dose acetylsalicylic acid (ASA) (OR 4), BMI ≤26 Kg/m2 (OR 4.1) and faecal calprotectin >500 µg/g (OR 5.5). A new score was developed using the variables mentioned above with an AUC of 0.86 (p<0.001 vs. Kane and Cotter scores). A score >10 had a sensitivity of 61.5% and a specificity of 92%. A score >17 gave a specificity of 100% with a sensitivity of 36%. The score was internally validated using bootstrapping techniques.

Although promising, the new scoring system must be externally validated before generalizing its use in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or older.
* Patient with chronic non-bloody watery diarrhoea (Bristol scale=6 or 7), with 2 or more liquid stools per day, of frequent occurrence (at least 3 times per week), of at least 1 month's duration.
* Normal blood test and biochemistry (including C reactive protein and TSH), negative anti-transglutaminase antibodies, and negative faecal ova and parasites. A 75SeHCAT is not mandatory.
* Patients with an indication for a diagnostic colonoscopy by their physician at charge, mainly to rule out MC.
* Signature of the study informed consent

Exclusion Criteria:

* Patients with either alternating diarrhoea-constipation or self-limiting diarrhoea at the time of colonoscopy.
* History of inflammatory bowel disease or coeliac disease, bile acid diarrhoea.
* Previous gastrointestinal surgery (excluding appendectomy or inguinal herniorrhaphy).
* Incomplete colonoscopy or no colon biopsies of at least right and left colon in separate containers (minimum 2 samples of each segment).
* Unsatisfactory preparation for a complete exploration (Boston scale <6, any segment <2)
* Significant macroscopic lesions on colonoscopy, other than those occasionally described in MC
* Inability to understand the instructions for participating in the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients derived at the digestive system department with chronic watery diarrhoea and clinical suspicion of MC, requiring colonoscopy with biopsies to complete the study
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients diagnosed with Microscopic Colitis (MC) | up to 2 months (after clinical and histological assessment)
  MC diagnosis based on clinical and histological criteria as established by the European guidelines on microscopic colitis: Miehlke S, Guagnozzi D, Zabana Y, et al. European guidelines on microscopic colitis: United European Gastroenterology and European Microscopic Colitis Group statements and recommendations [published online ahead of print, 2021 Feb 22]. United European Gastroenterol J. 2021;9(1):13-37

SECONDARY OUTCOMES:
Faecal calprotectin concentration (μg/g) | at inclusion (prior to colonoscopy)
  Faecal calprotectin concentration (μg/g) will be measured using a DSX system analyser (Dynex technologies, Worthing, UK) by ELISA (BÜHLMANN fCAL, Schönenbuch, Switzerland or similar)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari MútuaTerrassa, Terrassa, Barcelona, Spain

REFERENCES:
- [Background] Miehlke S, Guagnozzi D, Zabana Y, Tontini GE, Kanstrup Fiehn AM, Wildt S, Bohr J, Bonderup O, Bouma G, D'Amato M, Heiberg Engel PJ, Fernandez-Banares F, Macaigne G, Hjortswang H, Hultgren-Hornquist E, Koulaouzidis A, Kupcinskas J, Landolfi S, Latella G, Lucendo A, Lyutakov I, Madisch A, Magro F, Marlicz W, Mihaly E, Munck LK, Ostvik AE, Patai AV, Penchev P, Skonieczna-Zydecka K, Verhaegh B, Munch A. European guidelines on microscopic colitis: United European Gastroenterology and European Microscopic Colitis Group statements and recommendations. United European Gastroenterol J. 2021 Feb 22;9(1):13-37. doi: 10.1177/2050640620951905. Online ahead of print. PMID 33619914
- [Background] Beaugerie L, Pardi DS. Review article: drug-induced microscopic colitis - proposal for a scoring system and review of the literature. Aliment Pharmacol Ther. 2005 Aug 15;22(4):277-84. doi: 10.1111/j.1365-2036.2005.02561.x. PMID 16097993
- [Background] Larsson JK, Sjoberg K, Vigren L, Benoni C, Toth E, Olesen M. Chronic non-bloody diarrhoea: a prospective study in Malmo, Sweden, with focus on microscopic colitis. BMC Res Notes. 2014 Apr 14;7:236. doi: 10.1186/1756-0500-7-236. PMID 24731750
- [Background] Fernandez-Banares F, de Sousa MR, Salas A, Beltran B, Piqueras M, Iglesias E, Gisbert JP, Lobo B, Puig-Divi V, Garcia-Planella E, Ordas I, Andreu M, Calvo M, Montoro M, Esteve M, Viver JM; RECOMINA Project, GETECCU Grupo Espanol de Enfermedades de Crohn y Colitis Ulcerosa. Epidemiological risk factors in microscopic colitis: a prospective case-control study. Inflamm Bowel Dis. 2013 Feb;19(2):411-7. doi: 10.1002/ibd.23009. PMID 23344243
- [Background] Kane JS, Rotimi O, Everett SM, Samji S, Michelotti F, Ford AC. Development and validation of a scoring system to identify patients with microscopic colitis. Clin Gastroenterol Hepatol. 2015 Jun;13(6):1125-31. doi: 10.1016/j.cgh.2014.12.035. Epub 2015 Jan 20. PMID 25616029
- [Background] Kane JS, Sood R, Law GR, Gracie DJ, To N, Gold MJ, Ford AC. Validation and modification of a diagnostic scoring system to predict microscopic colitis. Scand J Gastroenterol. 2016 Oct;51(10):1206-12. doi: 10.1080/00365521.2016.1186221. Epub 2016 May 31. PMID 27243102
- [Background] Cotter TG, Binder M, Harper EP, Smyrk TC, Pardi DS. Optimization of a Scoring System to Predict Microscopic Colitis in a Cohort of Patients With Chronic Diarrhea. J Clin Gastroenterol. 2017 Mar;51(3):228-234. doi: 10.1097/MCG.0000000000000565. PMID 27404403
- [Background] Fernandez-Banares F, Casanova MJ, Arguedas Y, Beltran B, Busquets D, Fernandez JM, Fernandez-Salazar L, Garcia-Planella E, Guagnozzi D, Lucendo AJ, Mancenido N, Marin-Jimenez I, Montoro M, Piqueras M, Robles V, Ruiz-Cerulla A, Gisbert JP; Spanish Microscopic Colitis Group (SMCG). Current concepts on microscopic colitis: evidence-based statements and recommendations of the Spanish Microscopic Colitis Group. Aliment Pharmacol Ther. 2016 Feb;43(3):400-26. doi: 10.1111/apt.13477. Epub 2015 Nov 24. PMID 26597122
- [Background] Limburg PJ, Ahlquist DA, Sandborn WJ, Mahoney DW, Devens ME, Harrington JJ, Zinsmeister AR. Fecal calprotectin levels predict colorectal inflammation among patients with chronic diarrhea referred for colonoscopy. Am J Gastroenterol. 2000 Oct;95(10):2831-7. doi: 10.1111/j.1572-0241.2000.03194.x. PMID 11051356
- [Background] Wildt S, Nordgaard-Lassen I, Bendtsen F, Rumessen JJ. Metabolic and inflammatory faecal markers in collagenous colitis. Eur J Gastroenterol Hepatol. 2007 Jul;19(7):567-74. doi: 10.1097/MEG.0b013e328058ed76. PMID 17556903
- [Background] Wagner M, Peterson CG, Stolt I, Sangfelt P, Agnarsdottir M, Lampinen M, Carlson M. Fecal eosinophil cationic protein as a marker of active disease and treatment outcome in collagenous colitis: a pilot study. Scand J Gastroenterol. 2011 Jul;46(7-8):849-54. doi: 10.3109/00365521.2011.571707. Epub 2011 May 11. PMID 21557718
- [Background] Stoicescu A, Becheanu G, Dumbrava M, Gheorghe C, Diculescu M. Microscopic colitis - a missed diagnosis in diarrhea-predominant irritable bowel syndrome. Maedica (Bucur). 2012 Jan;7(1):3-9. PMID 23118812
- [Background] Batista L, Ruiz L, Ferrer C, Zabana Y, Aceituno M, Arau B, Andujar X, Esteve M, Fernandez-Banares F. Usefulness of fecal calprotectin as a biomarker of microscopic colitis in a cohort of patients with chronic watery diarrhoea of functional characteristics. Dig Liver Dis. 2019 Dec;51(12):1646-1651. doi: 10.1016/j.dld.2019.07.002. Epub 2019 Aug 2. PMID 31383457
- [Background] Palsson OS, Whitehead W, Tornblom H, Sperber AD, Simren M. Prevalence of Rome IV Functional Bowel Disorders Among Adults in the United States, Canada, and the United Kingdom. Gastroenterology. 2020 Apr;158(5):1262-1273.e3. doi: 10.1053/j.gastro.2019.12.021. Epub 2020 Jan 7. PMID 31917991
- [Background] Legrand E. Aceclofenac in the management of inflammatory pain. Expert Opin Pharmacother. 2004 Jun;5(6):1347-57. doi: 10.1517/14656566.5.6.1347. PMID 15163279
- [Background] Lanas A. Nonsteroidal antiinflammatory drugs and cyclooxygenase inhibition in the gastrointestinal tract: a trip from peptic ulcer to colon cancer. Am J Med Sci. 2009 Aug;338(2):96-106. doi: 10.1097/MAJ.0b013e3181ad8cd3. PMID 19680014
- [Background] Sandler RS, Keku TO, Woosley JT, Sandler DP, Galanko JA, Peery AF. Obesity is associated with decreased risk of microscopic colitis in women. World J Gastroenterol. 2022 Jan 14;28(2):230-241. doi: 10.3748/wjg.v28.i2.230. PMID 35110947